CLINICAL TRIAL: NCT00239538
Title: Prospective, Randomized, Open-label, Blinded Endpoint, Forced Titration Study to Compare Telmisartan Combined With HCTZ (80mg/12.5mg), to Valsartan Combined With HCTZ (160mg/12.5mg), for the Control of Mild-to-moderate Hypertension in Obese Patients With Type 2 Diabetes Mellitus Using ABPM.
Brief Title: SMOOTH - Blood Pressure Control in Diabetic/Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.399
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Hydrochlorothiazide

INTERVENTIONS:
Drug: telmisartan combined with hydrochlorothiazide (80/12.5 mg)
Drug: valsartan combined with hydrochlorothiazide (160/12.5mg)

SUMMARY:
The primary objective of this study is to demonstrate that telmisartan 80 mg combined with hydrochlorothiazide 12.5 mg (T80/H12.5) is at least as effective and possibly superior to valsartan 160 mg combined with hydrochlorothiazide 12.5 mg (V160/H12.5) in lowering mean ambulatory systolic blood pressure (SBP) and diastolic blood pressure (DBP) during the last 6 hours of the 24-hour dosing interval at the end of a 10-week treatment period in mild-to-moderate hypertensive, overweight or obese patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
Methodology:

Prospective, randomised, open-label, blinded end-point, forced-titration, parallel group comparison using Ambulatory Blood Pressure Monitoring (ABPM).

Planned/Actual Number of Subjects:

Enrolled: 1500/2085; Randomised: 750/840; Complete: 680/752

Diagnosis and Main Criteria for Inclusion:

1) Mild-to-moderate hypertension defined as a baseline mean seated cuff DBP of 95 - 109 (inclusive) mmHg, and/or SBP of 140-179 (inclusive) mmHg, and a baseline 24-hour ABPM mean DBP >= 85 mmHg, and/or SBP >= 130 mmHg. 2) Overweight or obese as defined by a Body Mass Index (BMI) >= 27 kg/m2 in non-Asians and >= 24 kg/m2 in Asians 3) Type-2 diabetes mellitus. 4) At least 30 years of age.

Duration of Treatment:

10 weeks total: telmisartan (80 mg) or valsartan (160 mg) for 4 weeks followed by telmisartan (80 mg) plus hydrochlorothiazide (12.5 mg) or valsartan (160 mg) plus hydrochlorothiazide (12.5 mg) for an additional 6 weeks.

Criteria for Efficacy:

Primary Endpoint:

Reductions in blood pressure during the last 6 hours of the 24-hour dosing interval as measured by ABPM. The primary analysis will consist of comparing telmisartan combined with hydrochlorothiazide 80 mg/12.5 mg to valsartan combined with hydrochlorothiazide 160 mg/12.5 mg at the end of the 10-week study using a closed testing procedure first testing for non-inferiority based on SBP; if significant, testing for non-inferiority based on DBP; if significant, testing for superiority based on SBP; and if significant, testing for superiority based on DBP.

Secondary Endpoints:

Statistically greater reductions in ambulatory blood pressure for patients treated with telmisartan combined with hydrochlorothiazide 80 mg/12.5 mg compared to patients treated with valsartan combined with hydrochlorothiazide 160 mg/12.5 mg at the end of the 10-week study as measured by: 1) Changes from baseline in the last 6 hours of the 24-hour dosing interval for pulse pressure; 2) Changes from baseline in the 24-hour ABPM mean (relative to dose time) for SBP, DBP, and pulse pressure; 3) Changes from baseline in the ABPM mean SBP, DBP, and pulse pressure (relative to clock time) during other periods (i.e., morning, daytime, night time) of the 24-hour dosing interval; 4) Change from baseline in systolic and diastolic blood pressure load during the 24-hour dosing interval; and 5) Percentage of patients responding to treatment based on the 24-hour ABPM mean SBP and DBP (relative to dose time).

Statistically greater reduction in mean seated trough blood pressure patients treated with telmisartan combined with hydrochlorothiazide 80 mg/12.5 mg compared to patients treated with valsartan combined with hydrochlorothiazide 160 mg/12.5 mg at the end of the 10-week study as measured by: 1) Changes from baseline in mean seated trough SBP and DBP as determined by electronic or manual device in-clinic; and 2) Percentage of patients responding to treatment based on electronic or manual in-clinic trough cuff blood pressures.

Evaluation of other endpoints comparing telmisartan combined with hydrochlorothiazide 80 mg/12.5 mg to valsartan combined with hydrochlorothiazide 160 mg/12.5 mg, respectively, including: 1) Changes from baseline in metabolic markers: serum TG, LDL-C, HDL-C, total cholesterol, potassium, fasting glucose and HbA1C, and for urine: Na, K, Cl, proteinuria (as measured by spot urine for protein:creatinine ratio); and 2) inflammatory markers: serum high sensitive C-reactive protein, serum homocysteine and plasma fibrinogen.

Criteria for Safety:

Evaluation of adverse events, physical examinations, laboratory assessments, pulse rate and cuff blood pressure monitoring.

Statistical Method:

Analysis of covariance with treatment and centre as main effects and baseline as a covariate; Mantel-Haenszel test controlling for centre.

Study Hypothesis:

Null Hypothesis:

The overall mean change from baseline in the automated blood pressure monitor mean blood pressure during the last 6 hours of the 24-hour dosing interval for telmisartan (80 mg) plus hydrochlorothiazide (12.5 mg) is less than or equal to that for valsartan (160 mg) plus hydrochlorothiazide (12.5 mg).

Alternative Hypothesis:

The overall mean change from baseline in the automated blood pressure monitor mean blood pressure during the last 6 hours of the 24-hour dosing interval for telmisartan (80 mg) plus hydrochlorothiazide (12.5 mg) is greater than that for valsartan (160 mg) plus hydrochlorothiazide (12.5 mg).

Comparison(s):

Telmisartan (80 mg) plus hydrochlorothiazide (12.5 mg) vs. valsartan (160 mg) plus hydrochlorothiazide (12.5 mg)

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Hypertension defined as a mean seated DBP of 95-109 (inclusive) mmHg, and/or SBP of 140-179 (inclusive) mmHg, measured by BpTRU electronic or manual cuff at Visit 2.
3. 24-hour mean DBP of >= 85 mmHg, and/or SBP = 130 mmHg, measured by ABPM at Visit 3.
4. 30 years of age or greater.
5. Ability to stop current antihypertensive therapy and other disallowed medications without risk to the patient.
6. Diagnosis of type-2 diabetes mellitus with HbA1C less than or equal to 10%.
7. Overweight or obese as defined by a BMI >= 27 kg/m2 in non-Asians and >= 24 kg/m2 in Asians.
8. Negative UPT for females.

Exclusion Criteria:

1. Pre-menopausal women, not surgically sterile or, not nursing/pregnant or are of child-bearing potential and will not practice acceptable methods of birth control during study.
2. Night shift workers
3. Mean sitting SBP >= 180 mmHg or mean sitting DBP >= 110 mmHg during any visit of the placebo run-in period.
4. Known or suspected secondary hypertension. Hepatic and/or renal dysfunction
5. Fasting serum glucose > 17 mmol/l (or 300 mg/dl) at visit 2
6. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, patients on dialysis or post-renal transplant patients.
7. Clinically relevant sodium depletion, hypokalaemia or hyperkalaemia.
8. Uncorrected volume depletion.
9. Primary aldosteronism.
10. Hereditary fructose intolerance.
11. Biliary obstructive disorders (e.g., cholestasis).
12. Congestive heart failure
13. Stroke within the past six months.
14. Documented severe obstructive coronary artery disease.
15. Myocardial infarction, cardiac surgery or unstable angina within the past three months.
16. PCI (percutaneous coronary intervention) within the past three months or planned during trial period.
17. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias.
18. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve.
19. Patients with type-1 diabetes mellitus.
20. Patients who have previously experienced symptoms of angioedema during ACE or ARB treatment.
21. History of drug or alcohol dependency in past six months.
22. Chronic administration of any medications known to affect blood pressure, except medication allowed by the protocol.
23. Any investigational drug therapy within the past month.
24. Known hypersensitivity to any component of the study drug.
25. Concurrent use of corticosteroids, colestipol or cholestyramine resins.
26. Any clinical condition which would not allow safe completion of the protocol.
27. Inability to comply with the protocol.
28. Any surgery that is, at the time of screening, planned to take place during the study period.
29. History of non-compliance with prescribed medications.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2003-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12

PRIMARY OUTCOMES:
Changes from baseline in the mean SBP and DBP as measured by ambulatory blood pressure monitoring (ABPM) | 10 weeks

SECONDARY OUTCOMES:
Changes from baseline in the last 6-hour ABPM mean (relative to dose time) pulse pressure. | 10 weeks
Changes from baseline in the 24-hour ABPM mean (relative to dose time) for SBP, DBP and pulse pressure. | 10 weeks
Changes from baseline in the ABPM mean (relative to clock time) for SBP, DBP, and pulse pressure during the morning, daytime and night time periods of the 24-hour dosing interval. | 10 weeks
Changes from baseline in SBP and DBP load during the 24-hour dosing interval. | 10 weeks
Responder rates based on the 24-hour ABPM mean (relative to dose time) blood pressures defined | 10 weeks
In-clinic trough cuff blood pressure measures at the end of both a 4-week (Visit 4) treatment period and a 10-week (Visit 6) treatment period. | 4 weeks and 10 weeks
Responder rates based on the mean seated trough cuff measurements | 4 weeks and 10 weeks
Metabolic and inflammatory marker changes from baseline | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Canada Ltd.
Locations (95):
- United States (55):
  - Cooper Green Hospital, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - Memorial Research Medical Clinic, Long Beach, California
  - 1200, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 8615, Nuena Park, California
  - Boehringer Ingelheim Investigational Site, Orange, California
  - Boehringer Ingelheim Investigational Site, Sacramento, California
  - 595, San Francisco, California
  - 1805, Stockton, California
  - Boehringer Ingelheim Investigational Site, Torrance, California
  - 2311, Washington D.C., District of Columbia
  - Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 6448, Hollywood, Florida
  - Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - Attention: Larry I. Gilderman, D.O., Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Pinellas Park, Florida
  - Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - Herron Medical Center, Ltd., Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Orland Park, Illinois
  - Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - Boehringer Ingelheim Investigational Site, Shawnee, Kansas
  - Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 200, Baltimore, Maryland
  - Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 12401, St Louis, Missouri
  - Boehringer Ingelheim Investigational Site, Missoula, Montana
  - Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 3, Buffalo, New York
  - Comprehensive Clinical Research, Bina, North Carolina
  - Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - Boehringer Ingelheim Investigational Site, Marion, Ohio
  - Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - Boehringer Ingelheim Investigational Site, Portland, Oregon
  - Boehringer Ingelheim Investigational Site, Broomal, Pennsylvania
  - 6605, Bartlett, Tennessee
  - 108, Fayetteville, Tennessee
  - Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 7777, Dallas, Texas
  - Boehringer Ingelheim Investigational Site, El Paso, Texas
  - Team Research of Texas, Harker Heights, Texas
  - Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 420, Salt Lake City, Utah
  - 20901, Ettrick, Virginia
  - Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 5000, Miwaukee, Wisconsin
- Argentina (3):
  - Boehringer Ingelheim Investigational Site, BsAs
  - Boehringer Ingelheim Investigational Site, Coronel Suárez
  - Boehringer Ingelheim Investigational Site, Rosario, Santa Fe
- Australia (3):
  - Boehringer Ingelheim Investigational Site, Kippa-Ring, Queensland
  - Emeritus Research, Malvern, Victoria
  - Boehringer Ingelheim Investigational Site, Prahran, Victoria
- Canada (23):
  - Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Conquitlam, British Columbia
  - Dr. Hugh Tildesley, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, North York, Ontario
  - Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - Boehringer Ingelheim Investigational Site, Orléans, Ontario
  - Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - LMC Thornhill, Thornhill, Ontario
  - Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 91 Thomas-Chapais, Boucherville, Quebec
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Pavillon St. Sacrement, Sainte-Foy, Quebec
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - c/o Hemodynamics Offices, Saskatoon, Saskatchewan
- Mexico (5):
  - Boehringer Ingelheim Investigational Site, Col. Magdalena de Las Salinas
  - Boehringer Ingelheim Investigational Site, Col. Sección 16, México, D.F.
  - Boehringer Ingelheim Investigational Site, Colonia del Valle
  - Boehringer Ingelheim Investigational Site, Guadalajara, Jalisco
  - Boehringer Ingelheim Investigational Site, Zapopan, Jalisco
- New Zealand (2):
  - Boehringer Ingelheim Investigational Site, Auckland
  - 1st Floor Hagely Hostel, Christchurch
- South Korea (3):
  - Inje University Pusan Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Korea University Medical Center, Seoul
- National Taiwan University Hospital, Taipei, Taiwan